CLINICAL TRIAL: NCT03878342
Title: Prospective Study of Omission of Whole-breast Radiotherapy Following Breast-conserving Surgery in Patients With Very Low Risk Ductal Carcinoma in Situ of the Breast
Brief Title: Radiotherapy Omission in Low Risk Ductal in Situ Carcinoma Breast
Acronym: ROMANCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: The French National Cancer Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UC-0107/1803
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: DCIS; Breast Cancer; Low Risk DCIS; Breast Conserving Surgery; Radiotherapy Omission
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Active Comparator): two fractionation regimens will be allowed for whole-breast irradiation: 50 Gy in 25 fractions over 5 weeks or 40 Gy in 15 fractions over 3 weeks. The delivery of an additional dose to the tumour bed (boost) will be at the referring physician discretion, according to the guidelines
  Interventions: Radiation: Radiotherapy
- No Radiotherapy (Experimental): No Irradiation- Active surveillance
  Interventions: Other: No Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — two fractionation regimens will be allowed for whole-breast irradiation: 50 Gy in 25 fractions over 5 weeks or 40 Gy in 15 fractions over 3 weeks. The delivery of an additional dose to the tumour bed (boost) will be at the referring physician discretion, according to the guidelines
  Arms: Radiotherapy
Other: No Radiotherapy — No Irradiation- Active surveillance
  Arms: No Radiotherapy

SUMMARY:
Following breast-conserving surgery (BCS) for localized ductal carcinoma in situ (DCIS) of the breast, whole-breast irradiation (WBRT) is a standard of care, reducing the absolute rate of in-breast recurrences (IBR) by more than 15% at 10 years, from 28% without radiotherapy to 13 % with radiotherapy. Half of the recurrences occurred as invasive disease. Whereas in the comparative trials, WBRT did not impact on overall survival, survival of patients who recurred with invasive cancers was impaired in comparison to patients who did not recur, or to patients with DCIS-only recurrences.

Using criteria based on age, tumor size, nuclear grade, and margins status, several trials and cohort studies failed to identify subgroups of patients at low risk, who could be safely spared the need for WBRT. The Radiation Therapy Oncology Group (RTOG) DCIS trial included patients treated with BCS for low- or intermediate grade DCIS revealed by unifocal microcalcifications, size ≤25 mm, margins ≥3 mm, and no residual microcalcifications after surgery. The 5-year rates of IBR were 3.5 % without radiotherapy, versus 0.4 % with radiotherapy, and 6.7 % and 0.9 % at 7 years, respectively (p <0.001). Sixty percent of the patients received tamoxifen in both groups.

Several studies showed that the same molecular classes were identified in DCIS as in invasive cancers. Studies suggested that low proliferation, hormone receptors expression, and lack of ERBB2 amplification were associated with a low risk of IBR in patients not receiving radiotherapy. A combined signature was tested in the Eastern Cooperative Oncology Group (ECOG) trial, showing a 10% IBR rate at ten years in patients with a low-risk.

Identifying very low-risk DCIS, using biological markers in addition to the clinical and histological markers of low-risk DCIS, could help to select patients who could be safely avoided WBRT following BCS. It would avoid over-treatment in these women and could decrease the cost of management.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged ≥50 years,
2. ECOG performance status ≤2
3. Microcalcifications on pre-biopsy mammography, unifocal, ≤25 mm or opacity without microcalcifications and no clinical palpable tumour
4. Absence of suspicious residual microcalcifications either on post-biopsy/ preoperative localization mammography, or on post-operative mammography Note: if absence of residual microcalcifications on post-biopsy/pre-operative mammography, post-operative mammography is not mandatory;
5. Breast-conserving surgical excision;
6. Histologically proven DCIS of the breast without an invasive component; Note Incidental histological finding of DCIS lesions developed within a benign breast lesion as well as an association with classical lobular carcinoma in situ (LCIS) associated with the DCIS are accepted.
7. Free margins (≥2 mm), or free margins following re-excision;
8. Low or Intermediate nuclear grade; Note: In case of nuclear grade heterogeneity within the same sample or between the biopsy or the surgical specimen, the highest nuclear grade score will prevail.
9. Tumour tissue sample availability; Note: Surgical specimen is mandatory unless no residual disease on the surgical specimen. In this instance, the initial diagnosis biopsy is required.
10. Absence of extensive necrosis (≤30% of the lumen diameter);
11. Immunohistochemical characteristics of luminal A subtype: ER≥10 %, PR ≥20 %, HER2 negative (0/1+) or 2+ not amplified (confirmed by fluorescent in situ hybridization (FISH) or chromogenic in situ hybridization (CISH)), Ki67 <15%.
12. Patient willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits and examinations and including follow-up;
13. Written informed consent.
14. Affiliation to the French social security.

Exclusion Criteria:

1. Endocrine treatment for breast cancer.
2. Previous invasive breast cancer including contralateral breast cancer, either metachronous or synchronous
3. Previous DCIS except contralateral DCIS in complete and continuous remission for more than 5 years
4. Previous other cancers (except basal-cell, carcinoma in situ of the cervix or endometrium), not in complete and continuous remission for more than 10 years
5. Known breast-cancer predisposing germ-cell mutation;
6. Palpable tumour with a diagnosis of DCIS on biopsy
7. Bloody nipple discharge;
8. Histological size >25 mm in one or multiple foci
9. High nuclear grade, including high nuclear grade in heterogeneous tumours;either on biopsy or on surgical specimen
10. Associated microinvasive or invasive component;
11. Presence of tumour cells in lymph nodes detected using H&E or immunohistochemical examination (if lymph node sentinel biopsy or dissection has been performed);
12. Absolute contra-indication to whole-breast irradiation as determined by the referring physician;
13. Patient unable to comply with study obligations for geographic, social, or physical reasons, or who is unable to understand the purpose and procedures of the study.
14. Pregnant women or breast feeding mothers,

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2029-11-14 (Estimated); Study Completion 2034-11-14 (Estimated)

PRIMARY OUTCOMES:
5-year cumulative incidence of in-breast cancer recurrences | 5 years
  Incidence of breast recurrence is determined from the date of last surgery to the date of breast recurrence.

SECONDARY OUTCOMES:
Overall survival (OS) | 10 years
  OS is defined as the interval between the date of last surgery and the date of death from any cause;
Breast cancer-specific survival (BCSS) | 10 years
  BCSS is defined as the interval between the date of last surgery and the date of death from breast cancer
Relapse-free survival (RFS) | 10 years
  RFS is defined as the interval between the date of last surgery and the date of ipsilateral breast recurrence, regional nodes recurrence, distant metastases, of death from breast cancer, whichever occurs first
Rate of in-breast recurrences (IBR). | 10 years
  In-breast recurrence defined as any carcinoma (invasive or in situ) occurring in the treated breast
Rate of Contralateral breast | 10 years
  Contralateral breast cancer defined as any carcinoma (invasive or in situ) occurring in the contralateral breast.
Quality of life of the patients using EORTC-QLQ-C 30 | 3 years
  Quality of life will be assessed using QLQ-C 30 questionnaire from the European Organization for Research and Treatment of Cancer (EORTC). It is a 30-item self-reporting questionnaire developed to assess the quality of life of cancer patients. It is grouped into five functional subscales (role, physical, cognitive, emotional and social functioning). In addition, there are three multi-item symptom scales (fatigue, pain, and nausea and vomiting), individual questions concerning common symptoms in cancer patients,and two questions assessing overall Quality of Life
Quality of life of the patients using EORTC-QLQ-BR23 | 3 years
  Quality of Life of Patients will be assessed using a EORTC-QLQ BR23.It is a 23-item self-reporting specific questionnaire developed to assess the quality of life of breast cancer patients. It permits to evaluate the symptoms of breast cancer and the side effects of treatment.
Cosmetics Evaluation | 3 years
  cosmetic results will be evaluated by centralized photographic analysis.
Long term toxicities | Throughout study completion, up to 10 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders and so the late effects and sequelea regarding the whole-breast radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alain FOURQUET, MD, Principal Investigator — Institut Curie
Locations (37):
- France (37):
  - Institut de Cancérologie de l'Ouest -Site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre d'Oncologie et de Radiothérapie du Pays Basque, Bayonne
  - Clinique Belharra, Bayonne
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier du Cotentin, Cherbourg
  - Centre Jean Perrin, Clermont-Ferrand
  - CHIC Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - Centre Georges Francois Leclerc, Dijon
  - Centre Hospitalier De Lagny Sur Marne, Jossigny
  - CHU Saint-Pierre La Réunion, La Réunion
  - Centre Guillaume le Conquérant, Le Havre
  - Centre Oscar Lambret, Lille
  - Chu De Limoges - Hopital Dupuytren, Limoges
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre de Radiothérapie Mermoz, Lyon
  - Centre Léon Berard, Lyon
  - Hôpital La Croix Rousse, Lyon
  - Institut Regional Du Cancer Montpellier Val D Aurelle, Montpellier
  - Centre Azuréen De Cancérologie, Mougins
  - Centre Antoine Lacassagne, Nice
  - Centre de Haute Energie, Nice
  - Hopital Pitie Salpetriere, Paris
  - Institut CURIE, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Frédéric Joliot, Rouen
  - Hôpital René Huguenin - Institut Curie, Saint-Cloud
  - CHU Saint-Etienne, Saint-Etienne
  - Centre De Radiothérapie De La Robertsau, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut De Cancerologie De Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No